CLINICAL TRIAL: NCT06692205
Title: Exploring the Effects of Primary Open-Angle Glaucoma on Visual-Motor Coordination
Brief Title: Effects of Primary Open-angle Glaucoma on Visual-motor Coordination
Status: Recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024KYPJ028
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-04

CONDITIONS: Primary Open-angle Glaucoma
Keywords: Visual-motor coordination; glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary open-angle glaucoma: Patients with primary open-angle glaucoma diagnosed by glaucoma professionals
- Healthy controls: Healthy controls were required to have a presenting Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity of 20/40 or better in both eyes.

SUMMARY:
Commonly used visual function assessments in glaucoma diagnosis and treatment-such as visual acuity, visual field, and contrast sensitivity-do not directly capture the impact of the disease on patients' daily abilities. While questionnaires can evaluate this impact from the patient's perspective, they are subject to individual biases and inconsistent evaluation standards. Thus, objective methods are needed to assess patients' abilities in visually guided daily activities. Grasping objects and avoiding obstacles are fundamental visually guided tasks that require effective visuomotor coordination. By attaching lightweight reflective markers to participants' limbs and using a motion capture system to track their movements in three-dimensional space, various indicators of planning, execution, and control in tasks such as object grasping and obstacle avoidance can be quantified, allowing for an objective evaluation of visuomotor coordination. However, it remains unclear how visuomotor coordination is affected in glaucoma patients at different disease stages or whether visual field damage in specific areas has distinct impacts on visuomotor coordination. This study, therefore, aims to investigate changes in visuomotor coordination among patients with primary open-angle glaucoma across disease stages and to determine the effects of visual field defects in different locations on their visuomotor abilities.

DETAILED DESCRIPTION:
Glaucoma is the leading cause of irreversible blindness worldwide, with an estimated 110 million glaucoma patients expected globally among individuals aged 40-80 by 2040. As a chronic and progressive eye disease, glaucoma can cause significant impairments in visual function. These impairments can severely limit daily activities like searching, walking, and reading, leading to a significant decline in patients' vision-related quality of life. Evaluating the visual abilities of glaucoma patients can not only gauge the extent of the disease's impact on their visual function but also indicate the effectiveness of clinical treatments and rehabilitation strategies. However, commonly used clinical tests, such as visual acuity and visual field, only partially reflect visual function and do not directly measure the disease's impact on daily activities. Questionnaires can be designed to assess the impact of the disease on daily activities, from the patient's perspective. However, as a subjective assessment method, questionnaires are susceptible to individual biases and evaluation standards. Therefore, more objective methods are needed to evaluate patients' performance and abilities in executing daily visually guided activities.

Grasping objects and avoiding obstacles are fundamental visually guided activities that require good visuomotor coordination. The visual system supplies essential information about the spatial position and intrinsic properties of objects, while the brain integrates this information to guide and control limb movements for specific tasks. By attaching lightweight reflective markers, such as spheres or patches, to participants' limbs and using a motion capture system to track these markers in three-dimensional space, various indicators of planning, execution, and control during tasks can be quantified. This approach enables an objective assessment of participants' visuomotor coordination abilities.

Previous studies have shown that glaucoma patients differ from age-matched healthy controls in reaching-grasping tasks, though findings on these differences have been inconsistent. Furthermore, researchers have reported that glaucoma patients also face challenges with mobility. However, it remains unclear how visuomotor coordination in glaucoma patients is affected across different disease stages during tasks like object grasping and obstacle avoidance, or whether the location of visual field damage has varied effects on their visuomotor coordination. In this study, we aim to compare the performance of patients with primary open-angle glaucoma and age-matched healthy controls in reaching-grasping and mobility tasks. Our goal is to investigate changes in visuomotor coordination across different stages of the disease and to clarify how visual field defects in various locations impact patients' visuomotor abilities.

ELIGIBILITY:
Inclusion Criteria:

1.1 Inclusion criteria of primary open-angle glaucoma group:

1. Age between 18 and 75 years;
2. Diagnosed with primary open-angle glaucoma, with no anti-glaucoma surgery scheduled within ±1 month;
3. Best corrected visual acuity in one eye ≥ 6/12;
4. Stereoscopic vision ≥ 1000 seconds of arc;
5. Able to clearly communicate and cooperate with the completion of relevant assessments and data collection.

1.2 Inclusion criteria of healthy controls：

1. Age between 18 and 75 years;
2. No history of eye disease other than refractive error and cataract;
3. Best corrected visual acuity in both eyes ≥ 6/12;
4. Stereoscopic vision ≥ 1000 seconds of arc;
5. Able to clearly communicate and cooperate with the completion of relevant assessments and data collection.

Exclusion Criteria:

1.1 Exclusion criteria for primary open-angle glaucoma group:

1. Individuals with cognitive dysfunction, psychological dysfunction, hearing impairment, or other conditions that prevent normal communication;
2. Presence of physical motor dysfunction, hyperthyroidism or hypothyroidism, malignant tumors, heart disease, or other systemic diseases;
3. Presence of other ocular conditions affecting visual function (except cataract and refractive error), such as age-related macular degeneration, diabetic retinopathy, optic neuropathy, retinal vascular disease, etc.;
4. Pregnant or lactating women.

1.2 Exclusion criteria for healthy controls：

1. Individuals with cognitive dysfunction, psychological dysfunction, hearing impairment, or other conditions that prevent normal communication;
2. Presence of physical motor dysfunction, hyperthyroidism or hypothyroidism, malignant tumors, heart disease, or other systemic diseases;
3. Presence of other ocular conditions affecting visual function (except cataract and refractive error), such as age-related macular degeneration, diabetic retinopathy, optic neuropathy, retinal vascular disease, etc.;
4. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Primary open-angle glaucoma: patients with primary open-angle glaucoma diagnosed by glaucoma professionals
  2. Healthy controls: subjects with no history of ocular disease, except for refractive errors and cataracts, and who have a presenting visual acuity of 20/40 or better in both eyes, as measured by the Early Treatment Diabetic Retinopathy Study (ETDRS) chart.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-21 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall movement duration of the reaching-and-grasping task | 1 day (Only once)
  Lightweight reflective markers are attached to the participants' thumb, index finger, and wrist joints, and a motion capture system is used to track the movement of these markers in three-dimensional space. The overall movement duration during the reaching-and-grasping task is then quantified. This overall movement duration serves as an index of task execution efficiency.
Overall movement duration of the mobility task | 1 day (Only once)]
  Lightweight reflective markers are attached to the participants' thigh, calf, and ankle joints, and a motion capture system is used to track the movement of these markers in three-dimensional space. The overall movement duration during the mobility task is then quantified, serving as an index of task execution efficiency during orientation and obstacle avoidance.

SECONDARY OUTCOMES:
ETDRS visual acuity | 1 day (Only once)]
  The information of Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity was obtained from the hospital electronic medical record system or outpatient medical record data.
Automatic perimetry report | 1 day (Only once)
  Automatic perimetry reports were obtained from the hospital electronic medical record system or outpatient medical record data. Mean defect (MD), mode standard deviation (PSD), corrected mode standard deviation (CPSD), short-term fluctuation (SF), glaucoma half field analysis (GHT), paracentric scotoma, nasal staircase, arch scotoma, tubular field and other characteristic visual field defects were recorded.
Pelli-Robson contrast sensitivity | 1 day (Only once)
  Pelli-Robson contrast sensitivity test card was used.
Stereoacuity | 1 day (Only once)
  Stereoacuity was measured using the Titmus stereopsis test.
Glaucoma Visual Functioning Questionnaire-40 (GVFQ-40) | 1 day (Only once)
  Glaucoma Visual Functioning Questionnaire-40 (GVFQ-40) is a 40-item questionnaire developed to evaluate the visual ability of glaucoma patients in detail. It consists of 40 items and measures the impact of glaucoma on restriction of participation in daily activities in five domains of functioning. Each item has six answer options, that is, no difficulty (score = 1), mild difficulty (score = 2), moderate difficulty (score = 3), extremely difficult (score = 4), completely unable to complete (score = 5), and do not perform for nonvisual reasons (no score). The GVFQ-40 is administered by a trained interviewer to all enrolled participants.
National Eye Institute-Visual Function Questionnaire-25 (NEI VFQ-25) | 1 day (Only once)
  The National Eye Institute-Visual Function Questionnaire-25 (NEI VFQ-25) is a valid and reliable vision-related quality of life (QOL) questionnaire designed for persons who have chronic eye diseases or low vision. It includes 25 items that comprise 11 subscales on different aspects of vision-related functioning and QOL and 1 item on general health. NEI VFQ-25 scores range from 0 to 100, with a higher score representing better functioning.
Short form 36 health survey questionnaire (SF-36) | 1 day (Only once)
  The Short Form 36 Health Survey Questionnaire (SF-36) is an instrument designed to measure health perception in a general population. It consists of 36 items and typically takes about five minutes to complete. The questionnaire assesses health across eight multi-item dimensions, covering functional status, well-being, and overall health evaluation. In six of the eight dimensions, patients are asked to rate their responses on three- or six-point scales. For each dimension, item scores are coded, summed, and transformed onto a scale ranging from 0 (worst health) to 100 (best health).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Opthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azoulay-Sebban L, Zhao Z, Zenouda A, Lombardi M, Gutman E, Brasnu E, Hamard P, Sahel JA, Baudouin C, Labbe A. Correlations Between Subjective Evaluation of Quality of Life, Visual Field Loss, and Performance in Simulated Activities of Daily Living in Glaucoma Patients. J Glaucoma. 2020 Oct;29(10):970-974. doi: 10.1097/IJG.0000000000001597. PMID 32649451
- [Background] Corveleyn X, Lenoble Q, Rouland JF, Boucart M. What is the Nature of the Reach-and-Grasp Deficit in Glaucoma? J Glaucoma. 2020 Sep;29(9):799-806. doi: 10.1097/IJG.0000000000001555. PMID 32858724
- [Background] Turano KA, Rubin GS, Quigley HA. Mobility performance in glaucoma. Invest Ophthalmol Vis Sci. 1999 Nov;40(12):2803-9. PMID 10549639
- [Background] Kotecha A, O'Leary N, Melmoth D, Grant S, Crabb DP. The functional consequences of glaucoma for eye-hand coordination. Invest Ophthalmol Vis Sci. 2009 Jan;50(1):203-13. doi: 10.1167/iovs.08-2496. Epub 2008 Sep 20. PMID 18806294
- [Background] Sivaprasad S, Tschosik E, Kapre A, Varma R, Bressler NM, Kimel M, Dolan C, Silverman D. Reliability and Construct Validity of the NEI VFQ-25 in a Subset of Patients With Geographic Atrophy From the Phase 2 Mahalo Study. Am J Ophthalmol. 2018 Jun;190:1-8. doi: 10.1016/j.ajo.2018.03.006. Epub 2018 Mar 10. PMID 29530781
- [Background] Ramulu PY, van Landingham SW, Massof RW, Chan ES, Ferrucci L, Friedman DS. Fear of falling and visual field loss from glaucoma. Ophthalmology. 2012 Jul;119(7):1352-8. doi: 10.1016/j.ophtha.2012.01.037. Epub 2012 Apr 4. PMID 22480738
- [Background] Bambo MP, Ferrandez B, Guerri N, Fuertes I, Cameo B, Polo V, Larrosa JM, Garcia-Martin E. Evaluation of Contrast Sensitivity, Chromatic Vision, and Reading Ability in Patients with Primary Open Angle Glaucoma. J Ophthalmol. 2016;2016:7074016. doi: 10.1155/2016/7074016. Epub 2016 Oct 31. PMID 27872754
- [Background] Tham YC, Li X, Wong TY, Quigley HA, Aung T, Cheng CY. Global prevalence of glaucoma and projections of glaucoma burden through 2040: a systematic review and meta-analysis. Ophthalmology. 2014 Nov;121(11):2081-90. doi: 10.1016/j.ophtha.2014.05.013. Epub 2014 Jun 26. PMID 24974815